CLINICAL TRIAL: NCT05738473
Title: The Effects of Intrapartum Antibiotic Prophylaxis to Prevent Group B Streptococcal Early-onset Disease on Maternal Vaginal Microbiome, Intestinal Microbiome and Immunity of Offspring
Brief Title: Effects of IAP-EOGBSD on Maternal Vaginal Microbiome, Offspring's Gut Microbiome and Metabolites.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Zhongshan Bo Ai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMOH2101
Record Dates: First submitted 2023-01-18; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Microbiome, Human
Keywords: Microbiome,; maternal and offspring; healthy; whole genome sequencing of GBS strain.; GBS test by(Q-PCR)
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women colonized by Group B Streptococcus (GBS) and undergoing IAP: vaginal microbiome of pregnant women colonized by Group B Streptococcus (GBS)、Pregnant women undergoing IAP
  Interventions: Drug: antibiotic
- pregnant women does not colonized by Group B Streptococcus (GBS) and not undergoing IAP: Group B streptococcus (GBS) does not colonize the vaginal microbiome of pregnant women、Pregnant wome

INTERVENTIONS:
Drug: antibiotic — For pregnant women with GBS colonization, antibiotics are used to prevent infection
  Groups: pregnant women colonized by Group B Streptococcus (GBS) and undergoing IAP

SUMMARY:
In view of the current status of prevention and research on GBS disease in mothers and infants at home and abroad, this project intends to explore the characteristics of vaginal microbiota of GBS-colonized pregnant women in southern China, the impact of IAP prevention of GBS-EOD on vaginal flora, and the effect of IAP prevention of GBS-EOD on intestinal flora and immune production in offspring, so as to improve the ability to prevent and treat GBS-related diseases in mothers and infants and promote maternal and infant health.

DETAILED DESCRIPTION:
This project intends to explore the characteristics of vaginal microbiota of GBS-colonized pregnant women in southern China, the impact of IAP prevention of GBS-EOD on vaginal flora, and the effect of IAP prevention of GBS-EOD on intestinal flora and immune production in offspring, so as to improve the ability to prevent and treat GBS-related diseases in mothers and infants and promote maternal and infant health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women are 18 to 40 years;
* 35 to 41 weeks of pregnancy;
* Singleton pregnancy;
* Plan for vaginal delivery and postpartum care in the research hospital;
* Pregnant women who volunteered to participate in the study.

Exclusion Criteria:

* Have infectious diseases, serious infections and clinical diseases;
* Use of antibiotics in the past 2 weeks;
* Long-term use of drugs due to digestion, immunity, blood, chronic diseases;
* Sexual behavior, vaginal douching and topical medication within 24 hours before sampling;
* Any medical or non-medical condition that the investigator considers inappropriate to participate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Pregnant women are 18 to 40 years; 2. 35 to 41 weeks of pregnancy
Sampling Method: Probability Sample
Enrollment: 492 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal flora | The offspring are born on the 3rd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the gut microbiome of offspring.
Secretory IgA | The offspring are born on the 3rd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.
Calprotectin | The offspring are born on the 3rd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the cailprotectin of offspring.
Intestinal flora | The offspring are born on the 42nd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the gut microbiome of offspring.
Secretory IgA | The offspring are born on the 42nd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the secretory IgA of offspring.
Calprotectin | The offspring are born on the 42nd day after birth
  Analyze the effect of intrapartum antibiotics on the prevention of early-onset group B streptococcal diseases on the cailprotectin of offspring.

SECONDARY OUTCOMES:
The effect of IAP to prevent GBS-EOD. | Vaginal flora on days 3rd after delivery.
  Analyze the effect of IAP (intrapartum antibiotics prophylaxis) to prevent GBS-EOD on maternal vaginal microbiome.
The characteristics of vaginal microbiome of pregnant women. | Vaginal flora on days 3rd after delivery.
  Analyze the characteristics of vaginal microbiome of pregnant women colonized by Group B Streptococcus (GBS).
The effect of IAP to prevent GBS-EOD. | Vaginal flora on days 42nd after delivery.
  Analyze the effect of IAP (intrapartum antibiotics prophylaxis) to prevent GBS-EOD on maternal vaginal microbiome.
The characteristics of vaginal microbiome of pregnant women. | Vaginal flora on days 42nd after delivery.
  Analyze the characteristics of vaginal microbiome of pregnant women colonized by Group B Streptococcus (GBS).

CONTACTS AND LOCATIONS:
Overall Officials: Qian Wang, Study Chair — Southern Medical University, China
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China